CLINICAL TRIAL: NCT06278558
Title: Study of the Psychological Factors Influencing Post-traumatic Growth During Oncological Pathway
Brief Title: Psychological Factors Influencing Cancer Post-traumatic Growth
Acronym: CEMA-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valenciennes (Network)
Collaborators: Ligue contre le cancer, France (Other); Centre Oscar Lambret (Other); Centre de Cancérologie Les Dentellières (Unknown); Clinique Teissier (Unknown); Hôpital Saint Vincent de Paul, Lille (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-02-01
Record Dates: First submitted 2023-12-07; First posted 2024-02-26 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Cancer; Post-traumatic growth; Emotional competence; Emotional distress
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic; Psychiatrists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interviews with a psychologist/psychiatrist (Experimental): Implementation of an interview with a psychologist or psychiatrist following a telephone conversation with patients with no psychological follow-up and a high HADS score (≥11), at all stages of the study (start of chemotherapy T1, end of chemotherapy T2, 6 months after the end of chemotherapy).
  Interventions: Other: Interviews with a psychologist/psychiatrist

INTERVENTIONS:
Other: Interviews with a psychologist/psychiatrist — All patients with a high score (≥11) on the HADS anxiety and/or depressive symptoms scale and who are not already receiving known psychological treatment or treatment mentioned in the file will be contacted by telephone by the investigator or a qualified person designated by him/her in order to conduct a telephone interview with the patient and refer him/her to a psychologist or psychiatrist if necessary. The number and percentage of consultations with a psychologist or psychiatrist following this telephone interview will be calculated in order to highlight the benefits of such a practice (HADS assessment + telephone interview with +/- referral) for earlier and easier referral. Depending on the number of patients contacted, consideration may be given to testing the effect of this approach on post-traumatic development.

SUMMARY:
The study focuses on post-traumatic growth (positive changes linked to appreciation of life, personal strengths, social relationships...) in the context of different types of cancer and with a longitudinal approach to the care pathway. The aim of the study is to better understand whether psychological variables (emotional competence, psychological flexibility, psychological distress) and patients' care satisfaction, assessed at the start of the cancer treatment pathway, can influence their post-traumatic growth at the end of the chemotherapy protocol and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients in the initial phase of curative treatment for a 1st solid cancer
* At the start of neo-adjuvant or adjuvant chemotherapy (1st course or 2nd course)
* At less than 6 months from the initial diagnosis
* Patient having given written consent to participate in the study

Exclusion Criteria:

* Patients with a previous history of cancer
* Patients with incurable cancer progression, recurrence or relapse
* Metastatic, brain, hematological or skin cancer
* Patients who have difficulty understanding written French
* Patient psychologically or physically unable to answer questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic growth | T1 : At the beginning of chemotherapy
  Post-traumatic growth will be assessed using a 21-item self-report questionnaire and a Likert scale ranging from 0 (Not at all) to 4 (Totally), the Posttraumatic growth inventory (PTGI), which has been revalidated in French (Dubuy et al., 2022) in 4 dimensions: new direction for life (6 items), personal abilities (6 items), spiritual change (2 items) and relationships with others (7 items).
Post-traumatic growth | T2 : Up to 3 weeks after the end of chemotherapy
  Post-traumatic growth will be assessed using a 21-item self-report questionnaire and a Likert scale ranging from 0 (Not at all) to 4 (Totally), the Posttraumatic growth inventory (PTGI), which has been revalidated in French (Dubuy et al., 2022) in 4 dimensions: new direction for life (6 items), personal abilities (6 items), spiritual change (2 items) and relationships with others (7 items).
Post-traumatic growth | T3 : 6 months after the end of chemotherapy protocol
  Post-traumatic growth will be assessed using a 21-item self-report questionnaire and a Likert scale ranging from 0 (Not at all) to 4 (Totally), the Posttraumatic growth inventory (PTGI), which has been revalidated in French (Dubuy et al., 2022) in 4 dimensions: new direction for life (6 items), personal abilities (6 items), spiritual change (2 items) and relationships with others (7 items).

SECONDARY OUTCOMES:
Satisfaction of supportive care needs | T1 : At the beginning of chemotherapy
  Patients' satisfaction of supportive care needs are assessed using the Supportive Care Needs Survey (SCNS), validated in French (Brédart et al., 2012), comprising 34 items and 5 dimensions (Physical and daily life, psychological and emotional, sexuality, information, care system).
Satisfaction of supportive care needs | T2 : Up to 3 weeks after the end of chemotherapy
  Patients' satisfaction of supportive care needs are assessed using the Supportive Care Needs Survey (SCNS), validated in French (Brédart et al., 2012), comprising 34 items and 5 dimensions (Physical and daily life, psychological and emotional, sexuality, information, care system).
Satisfaction of supportive care needs | T3 : 6 months after the end of chemotherapy protocol
  Patients' satisfaction of supportive care needs are assessed using the Supportive Care Needs Survey (SCNS), validated in French (Brédart et al., 2012), comprising 34 items and 5 dimensions (Physical and daily life, psychological and emotional, sexuality, information, care system).
Emotional competence | T1 : At the beginning of chemotherapy
  Emotional competence are assessed using the Profile of Emotional Competence (S-PEC), validated in French (Baudry et al., 2020), comprising 13 items and 2 dimensions (intrapersonal and interpersonal emotional skills).
Emotional competence | T2 : Up to 3 weeks after the end of chemotherapy
  Emotional competence are assessed using the Profile of Emotional Competence (S-PEC), validated in French (Baudry et al., 2020), comprising 13 items and 2 dimensions (intrapersonal and interpersonal emotional skills).
Emotional competence | T3 : 6 months after the end of chemotherapy protocol
  Emotional competence are assessed using the Profile of Emotional Competence (S-PEC), validated in French (Baudry et al., 2020), comprising 13 items and 2 dimensions (intrapersonal and interpersonal emotional skills).
Anxiety and depression symptoms | T1 : At the beginning of chemotherapy
  Anxiety and depressive symptoms were assessed using the Hospital Anxiety and Depression Scale (HADS), validated in French (Razavi et al., 1989), comprising 14 items and 2 dimensions (anxiety and depression).
Anxiety and depression symptoms | T2 : Up to 3 weeks after the end of chemotherapy
  Anxiety and depressive symptoms were assessed using the Hospital Anxiety and Depression Scale (HADS), validated in French (Razavi et al., 1989), comprising 14 items and 2 dimensions (anxiety and depression).
Anxiety and depression symptoms | T3 : 6 months after the end of chemotherapy protocol
  Anxiety and depressive symptoms were assessed using the Hospital Anxiety and Depression Scale (HADS), validated in French (Razavi et al., 1989), comprising 14 items and 2 dimensions (anxiety and depression).
Psychological flexibility | T1 : At the beginning of chemotherapy
  Psychological flexibility is assessed using the multidimensional psychological flexibility inventory (MPFI-24), validated in French (Grégoire et al., 2020), consisting of 24 items and 2 dimensions (flexibility and inflexibility).
Psychological flexibility | T2 : Up to 3 weeks after the end of chemotherapy
  Psychological flexibility is assessed using the multidimensional psychological flexibility inventory (MPFI-24), validated in French (Grégoire et al., 2020), consisting of 24 items and 2 dimensions (flexibility and inflexibility).
Psychological flexibility | T3 : 6 months after the end of chemotherapy protocol
  Psychological flexibility is assessed using the multidimensional psychological flexibility inventory (MPFI-24), validated in French (Grégoire et al., 2020), consisting of 24 items and 2 dimensions (flexibility and inflexibility).

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Baudry, Principal Investigator — CH de Valenciennes
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, France

IPD SHARING:
Plan to Share IPD: No